CLINICAL TRIAL: NCT04759937
Title: Immunochromatography Versus Microscopy for Diagnosis of Entamoeba Histolytica/Dispar Infection in Sohag.
Brief Title: Immunochromatography Versus Microscopy for Diagnosis of Entamoeba Histolytica/Dispar Infection.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Khoulood Zakaria Hashem, Demonstrator at medical parasitology department, Faculty of medicine, Sohag University
Other Study IDs: Soh-Med-21-02-16
Record Dates: First submitted 2021-02-14; First posted 2021-02-18 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Dysentery Amebic
Keywords: dysentery; diarrhea; Entamoeba; histolytica; dispar
MeSH Terms: conditions — Amebiasis; Dysentery; Diarrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — stool specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Amoebiasis, an infection by the protozoan parasite Entamoeba histolytica is globally considered as the third leading parasitic cause of human mortality besides malaria and schistosomiasis. It is estimated that E. histolytica may infect half a billion people annually. Moreover, it was estimated that 100,000 patients per year died due to the clinical complications of the disease. Laboratory diagnosis of E. histolytica/dispar is usually achieved by microscopic detection of trophozoites or cysts in stool samples. Microscopy is time consuming and requires an experienced observer to identify the organism. Furthermore, it must be performed on three stool samples to increase sensitivity leading to decreased patient compliance and delay in the final diagnosis. Therefore, a few the commercially available copro-antigen assay have been developed for E. histolytica/dispar diagnosis including the enzyme immunoassay and non-enzymatic immunochromatographic (ICT) assays that do not depend on microscopy skills and increase laboratory efficiency by reducing time and cost.

The aim of the study is:

1. to evaluate the efficacy of commercially available rapid immunochromatographic Copro-antigen assay (RIDA® QUICK Entamoeba) in comparison with conventional microscopic examination for the diagnosis of E. histolytica /dispar infection.
2. to estimate the prevalence of E. histolytica /dispar infection in outpatients in Sohag.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of dysentery or diarrhea with any age & sex groups.

Exclusion Criteria:

* Patients taking amoebicidal drugs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: samples will be collected from outpatients complaining of dysentery or diarrhea with any age & sex groups from different locations (cities and village).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
evaluate the efficacy of immunochromatographic Copro-antigen assay for diagnosis of Entamoeba histolytica/ dispar. | 16 weeks following the startpoint of the study.
  comparing the sensitivity and specifity with conventional microscopy for diagnosis of Entamoeba histolytica/ dispar infection.

SECONDARY OUTCOMES:
detect the prevelance of Entamoeba histolytica/ dispar in Sohag. | 16 weeks following the startpoint of the study.
  By examining stool samples from 100 patients, the number of cases with Entamoena histolytica/dispar infection is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine-Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided